CLINICAL TRIAL: NCT01837108
Title: Effects of the Selective Mineralocorticoid Receptor Antagonist Eplerenone on Extracellular Adenosine Formation in Humans in Vivo
Brief Title: Eplerenone and Extracellular Adenosine Formation
Acronym: eplerenone01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NL43234.091.13
Record Dates: First submitted 2013-04-12; First posted 2013-04-22 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-04

CONDITIONS: Pharmacodynamics
Keywords: healthy
MeSH Terms: interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): fully mimicking placebo 50 mg bid during 8 days
  Interventions: Drug: Placebo
- eplerenone (Experimental): eplerenone 50 mg bid during 8 days
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — 2 tabs of eplerenone 25 mg will be over-encapsulated and a fully mimicking placebo will be provided by the department of clinical pharmacy of the Radboud University Medical Centre Nijmegen
  Other Names: Inspra, RVG 29963
  Arms: eplerenone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Various studies have reported cardioprotective effects of mineralocorticoid receptor (MR) antagonists in the setting of an acute myocardial infarction. In a recent animal study, the protective effect of MR antagonists on infarct size was completely abolished in CD73 knock-out and adenosine A2b receptor knock-out mice, and by co-administration of adenosine receptor antagonists in rats. These findings suggest that extracellular formation of adenosine is crucial for this protective effect and that MR antagonists stimulate extracellular adenosine formation by the enzyme CD73.

To investigate whether eplerenone promotes adenosine receptor stimulation by activating CD73, the investigators will measure forearm blood flow in response to various dosages of dipyridamole with the use of plethysmography. Dipyridamole increases the extracellular endogenous adenosine concentration by inhibition of the ENT transporter and induces local vasodilation. Therefore, the vasodilator effect of dipyridamole accurately reflects extracellular adenosine formation by the CD73 enzyme.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 18-40 years
* Healthy
* Written informed consent

Exclusion Criteria:

* Smoking
* Hypertension (Blood pressure >140 mmHg and/or >90 mmHg - SBP/DBP-)
* Hypotension (Blood pressure <100 mmHg and/or <60 mmHg -SBP/DBP-)
* Diabetes Mellitus (fasting glucose > 6.9 mmol/L or random > 11.0 mmol/L in venous plasma)
* History of any cardiovascular disease
* Angina pectoris
* History of chronic obstructive pulmonary disease (COPD) or asthma
* Alcohol and/or drug abuse
* Concomitant use of medication
* Renal dysfunction (MDRD < 60 ml/min/1.73 m2)
* Liver enzyme abnormalities (ALAT > twice upper limit of normality)
* Serum potassium ≥ 4.8 mmol/L
* Fasting total cholesterol > 6.0 mmol/L
* Second/third degree AV-block on electrocardiography

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
forearm blood flow response | 8 days
  Forearm blood flow response to the intrabrachial administration of incremental dosages of dipyridamole, after treatment with eplerenone, compared to placebo. The forearm blood flow will be measured by plethysmography.

SECONDARY OUTCOMES:
forearm blood flow | 8 days
  Forearm blood flow response to the intrabrachial administration of incremental dosages of dipyridamole, with and without caffeine, after eplerenone treatment. The forearm blood flow will be measured by plethysmography.
forearm blood flow | 8 days
  Forearm blood flow to incremental periods of arterial occlusion. The forearm blood flow will be measured by plethysmography.

OTHER OUTCOMES:
24 hours urine sample | 1 day
  Twenty-four hours urine samples will be collected and sodium and creatinine will be determined, to ensure that salt intake is approximately the same during both treatment days.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Riksen, Dr., Principal Investigator — Radboud University Medical Centre Nijmegen; Gerard Rongen, Prof., Study Chair — Radboud University Medical Centre Nijmegen
Locations (1):
- Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] van den Berg TN, Deinum J, Bilos A, Donders AR, Rongen GA, Riksen NP. The effect of eplerenone on adenosine formation in humans in vivo: a double-blinded randomised controlled study. PLoS One. 2014 Oct 30;9(10):e111248. doi: 10.1371/journal.pone.0111248. eCollection 2014. PMID 25356826